CLINICAL TRIAL: NCT01673711
Title: Correlation of [D10] Phenanthrene Metabolism With Bronchoepithelial Dysplasia and Metaplasia in Smokers at High Risk for Lung Cancer
Brief Title: Deuterated Phenanthrene Tetraol in Smokers Who Are at High Risk For Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2011NTUC092; NCI-2012-01148 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-02; First posted 2012-08-28 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer; Squamous Lung Dysplasia; Tobacco Use Disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder | interventions — phenanthrene

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood, buccal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basic Science (deuterated phenanthrene tetraol): Patients receive deuterated phenanthrene tetraol PO and collect urine for 6 hours after dosing.
  Interventions: Drug: deuterated phenanthrene tetraol; Drug: pharmacological study; Drug: laboratory biomarker analysis

INTERVENTIONS:
Drug: deuterated phenanthrene tetraol — Given PO
  Other Names: [D10] phenanthrene; phenanthrene-D10
Drug: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies deuterated phenanthrene tetraol in smokers who are at high risk for lung cancer. Studying samples of urine in the laboratory from smokers who are at high risk for lung cancer may help doctors learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relationship between urinary deuterated ([D10]) phenanthrene tetraol (PheT) level, PheT:phenanthrols (HOPhe) ratio, and the presence of bronchoepithelial metaplasia and/or dysplasia in smokers who have undergone screening bronchoscopy at Roswell Park Cancer Institute (RPCI).

OUTLINE:

Patients receive deuterated phenanthrene tetraol orally (PO). Urine samples are collected for laboratory studies for 6 hours after dosing.

ELIGIBILITY:
* Current or former smoker
* 18 years of age or older
* Documentation of a diagnosis of no dysplasia, dysplasia, or metaplasia on bronchoscopy (white light and/or autofluorescence) conducted less than or equal to 10 years prior to registration
* Not pregnant or breastfeeding
* Able to provide written informed consent indicating an understanding of the nature of the study
* Willing to comply with study requirements, including taking [D10]phenanthrene in water with 20% ethanol
* No previous history of aerodigestive cancer
* Not currently undergoing treatment for any cancers. Exception: basal cell or squamous cell skin cancer
* Not currently taking any other investigational agents
* No history of allergic reaction to [D10]phenanthrene or similar compounds
* No major medical comorbidities, for example, renal dysfunction, heart function, and diabetes, to be adjudicated by study physicians
* Not a former or recovering alcoholic
* No use of metronidazole or antabuse less than or equal to 7 days prior to [D10]phenanthrene dosing, as they could potentially interact with ethanol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy current and former smokers
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Urinary deuterated phenanthrene tetraol level | Up to 6 hours
  A multiple regression analysis will be performed including explanatory variables such as lesion status, presence/absence of chronic obstructive pulmonary disease (COPD) or asbestos, duration of smoking, smoking intensity, age, and gender.
PheT:HOPhe ratio | Up to 6 hours
  A multiple regression analysis will be performed including explanatory variables such as lesion status, presence/absence of COPD or asbestos, duration of smoking, smoking intensity, age, and gender.
Correlation of deuterated phenanthrene tetraol level and PheT:HOPhe ratio with the presence of bronchoepithelial metaplasia and/or dysplasia | Up to 6 hours
  A multiple regression analysis will be performed including explanatory variables such as lesion status, presence/absence of COPD or asbestos, duration of smoking, smoking intensity, age, and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Hecht, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
- BC Cancer Agency, Vancouver, British Columbia, Canada